CLINICAL TRIAL: NCT03738943
Title: Pyridoxine, P2 Receptor Antagonism, and ATP-mediated Vasodilation in Young Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Frank Dinenno, Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-7430H
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Receptor Blockade
Keywords: Adenosine Triphosphate; Pyridoxine; Cardiovascular; PLP; P5P
MeSH Terms: interventions — Adenosine Triphosphate; Acetylcholine; Nitroprusside; Adenosine Diphosphate; Adenosine Monophosphate; Uridine Triphosphate; Adenosine; Vitamin B 6; Pyridoxine; Pyridoxal Phosphate

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three arms of the study. The arms of the study are based on the vasodilators being tested in order to determine the effect of pyridoxine or PLP on vasodilation in response to intra-arterial administration of the vasodilators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ATP, Ach, SNP (Experimental): All drugs will be administered via intra-arterial (brachial artery) infusion, and the dosages below will be administered two times: once before administration of Vitamin B6 (pyridoxine) and once following administration of the Vitamin B6 (pyridoxine) loading dose.
  Adenosine Triphosphate: 1.25, 2.5, 5, and 10 μg/dl forearm volume/min for 3 minutes each.
  Acetylcholine: 1, 4, 8, and 16 μg/dl forearm volume/min for 3 minutes each.
  Sodium Nitroprusside: 0.25, 0.5, 1, and 2 μg/dl forearm volume/min for 3 minutes each.
  Vitamin B6 (pyridoxine): up to 200 mg of pyridoxine will be infused over 20 minutes. A maintenance dose of 2.5 mg/min may be used throughout the remainder of the protocol.
  Pyridoxal-5-Phosphate (PLP) may be used as an alternative blocker instead of pyridoxine. It will be infused at doses up to 200 µg/dl forearm volume/min.
  Interventions: Drug: Adenosine Triphosphate; Drug: Acetylcholine; Drug: Sodium Nitroprusside; Drug: Vitamin B 6; Drug: Pyridoxal 5'-Phosphate
- ATP, ADP, AMP (Experimental): All drugs will be administered via intra-arterial (brachial artery) infusion, and the dosages below will be administered two times: once before administration of Vitamin B6 (pyridoxine) and once following administration of the Vitamin B6 (pyridoxine) loading dose.
  Adenosine Triphosphate: 1.25, 2.5, 5, and 10 μg/dl forearm volume/min for 3 minutes each.
  Adenosine Diphosphate: 20, 40, 80, and 160 μg/dl forearm volume/min for 3 minutes each.
  Adenosine Monophosphate: 25, 50, 100, and 200 μg/dl forearm volume/min for 3 minutes each.
  Vitamin B6 (pyridoxine): up to 200 mg of pyridoxine will be infused over 20 minutes. A maintenance dose of 2.5 mg/min may be used throughout the remainder of the protocol.
  Pyridoxal-5-Phosphate (PLP) may be used as an alternative blocker instead of pyridoxine. It will be infused at doses up to 200 µg/dl forearm volume/min.
  Interventions: Drug: Adenosine Triphosphate; Drug: Adenosine Diphosphate; Drug: Adenosine Monophosphate; Drug: Vitamin B 6; Drug: Pyridoxal 5'-Phosphate
- ATP, UTP, Adenosine (Experimental): All drugs will be administered via intra-arterial (brachial artery) infusion, and the dosages below will be administered two times: once before administration of Vitamin B6 (pyridoxine) and once following administration of the Vitamin B6 (pyridoxine) loading dose.
  Adenosine Triphosphate: 1.25, 2.5, 5, and 10 μg/dl forearm volume/min for 3 minutes each.
  Uridine Triphosphate: 1.25, 2.5, 5, and 10 μg/dl forearm volume/min for 3 minutes each.
  Adenosine: 3.125, 6.25, 12.5, and 25 μg/dl forearm volume/min for 3 minutes each.
  Vitamin B6 (pyridoxine): up to 200 mg of pyridoxine will be infused over 20 minutes. A maintenance dose of 2.5 mg/min may be used throughout the remainder of the protocol.
  Pyridoxal-5-Phosphate (PLP) may be used as an alternative blocker instead of pyridoxine. It will be infused at doses up to 200 µg/dl forearm volume/min.
  Interventions: Drug: Adenosine Triphosphate; Drug: Uridine Triphosphate; Drug: Adenosine; Drug: Vitamin B 6; Drug: Pyridoxal 5'-Phosphate

INTERVENTIONS:
Drug: Adenosine Triphosphate — See arm/group descriptions
  Other Names: ATP
Drug: Acetylcholine — See arm/group descriptions
  Other Names: Ach
  Arms: ATP, Ach, SNP
Drug: Sodium Nitroprusside — See arm/group descriptions
  Other Names: SNP
  Arms: ATP, Ach, SNP
Drug: Adenosine Diphosphate — See arm/group descriptions
  Other Names: ADP
  Arms: ATP, ADP, AMP
Drug: Adenosine Monophosphate — See arm/group descriptions
  Other Names: AMP
  Arms: ATP, ADP, AMP
Drug: Uridine Triphosphate — See arm/group descriptions
  Other Names: UTP
  Arms: ATP, UTP, Adenosine
Drug: Adenosine — See arm/group descriptions
  Other Names: Adenocard
  Arms: ATP, UTP, Adenosine
Drug: Vitamin B 6 — See arm/group descriptions
  Other Names: Pyridoxine; Pyridoxine Hydrochloride
Drug: Pyridoxal 5'-Phosphate — See arm/group descriptions
  Other Names: PLP; P5P; pyridoxal phosphate monohydrate; MC-1

SUMMARY:
Previous research has identified adenosine triphosphate (ATP) as an important vasodilator that is released from red blood cells during exercise and exposure to hypoxic environments in adult humans. Further, older adults appear to have lower blood flow during both of these stressors and also have lower amounts of ATP released from their red blood cells. However, the contribution of ATP to vasodilation in response to exercise and hypoxia is currently unknown due to the lack of an effective ATP receptor antagonist. We aim to determine whether Vitamin B6 or its metabolite, Pyridoxal-5-Phosphate (PLP) is an effective ATP receptor antagonist.

DETAILED DESCRIPTION:
Adenosine triphosphate (ATP) is an established vasodilator that is released from red blood cells during a variety of stimuli including exercise and exposure to hypoxic environments. Many studies have shown that infusion of ATP can lead to vasodilation similar to that which is achieved during exercise, and that plasma ATP concentrations increase in a graded fashion during graded exercise. Further, older adults have lower levels of blood flow during exercise and hypoxia compared to their younger counterparts, and the reduced blood flow is coupled with impaired release of ATP from red blood cells during these stimuli. Thus, ATP is believed to be an important vasodilator. However, the role of ATP in the regulation of blood flow is not fully understood due to the lack of an effective ATP receptor (P2Y2) antagonist. Development of an effective P2Y2 antagonist will allow researchers to determine the role of ATP in vasodilation to stimuli such as exercise by comparing blood flow during exercise with and without the blocker. Preliminary data from our laboratory suggests that Vitamin B6 (pyridoxine hydrochloride) or its metabolite Pyridoxal-5-Phosphate (PLP) may be an effective blocker of ATP-mediated vasodilation. As a result, the purpose of this study is to determine whether Vitamin B6 or PLP can inhibit vasodilation in response to intra-arterial infusions of ATP. This study also aims to determine the specificity of Vitamin B6 or PLP by measuring its effect on vasodilation in response to infusion of several other vasodilators.

Participants will be asked to complete one screening visit and one study visit. Once study eligibility has been determined, participants will report to the Human Performance Clinical Research Laboratory at Colorado State University following an overnight fast. A physician will then place a catheter in the brachial artery of the non-dominant arm, and participants will be randomized into one of three study arms to determine which drugs will be infused into the artery. Each arm includes ATP and two other vasodilators. The study will begin by measuring vasodilation in response to four standard doses of each vasodilator. Vasodilation in response to the vasodilators will then be assessed again following infusion of Vitamin B6 or PLP. Reduced vasodilation to any of the drugs during the second trial will suggest that Vitamin B6 or PLP is an antagonist to the channel through which the drug signals. Each study visit will last approximately 4-5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary-moderately active
* Free of chronic disease

Exclusion Criteria:

* Current smoker
* BMI > 29.9 kg/m2
* Blood pressure equal to or greater than 140/90 mmHg
* Use of any medications including vitamin B6 supplements or antioxidants

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Vascular Conductance | Continuous measurement of vascular conductance during the 12 minute dose response for each drug. Measures are repeated following administration of Vitamin B6 or PLP.
  Vascular conductance is an index of vascular tone through which vasodilation can be determined. Vascular conductance is calculated by measuring blood flow in response to infusion of a vasodilator and accounting for blood pressure. Thus, the change in blood flow is due to a change in vascular conductance.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Dinenno, PhD, Principal Investigator — Colorado State University
Locations (1):
- Human Performance and Clinical Research Laboratory, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No